CLINICAL TRIAL: NCT01745380
Title: A Phase 3, Multi-Center, Randomized, Double-Blind, Parallel-Groups Clinical Trial Comparing the Efficacy and Safety of Intranasally Administered Kovacaine Mist to Placebo for Anesthetizing Maxillary Teeth in Adults
Brief Title: Comparison of Intranasal Kovacaine Mist, and Placebo for Anesthetizing Maxillary Teeth in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Renatus, LLC (Industry)
Collaborators: Triligent International (Industry); Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR 3-03
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Anesthesia
Keywords: operative; dental procedure
MeSH Terms: interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kovacaine Mist (Experimental): Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - 2 sprays will be administered at the start of the procedure, if anesthesia is insufficient, a third spray will be administered.
  Interventions: Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
- Placebo (Placebo Comparator): Placebo - 2 sprays will be administered at the start of the procedure, if anesthesia is insufficient, a third spray will be administered.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% — The study drug is regional anesthetic delivered intranasally on the same side as the operative tooth
  Other Names: Kovacaine Mist
  Arms: Kovacaine Mist
Drug: Placebo — The placebo spray was identical in appearance to and was administered in the same volume and manner as the active ingredient.
  Other Names: inactive ingredients
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy of Kovacaine Mist, and Placebo for inducing pulpal anesthesia of the maxillary teeth in adults.

DETAILED DESCRIPTION:
The study will employ a multi-center, randomized, double-blind, placebo-controlled, parallel-groups design to assess the safety and efficacy of Kovacaine Mist delivered intranasally for inducing pulpal anesthesia of maxillary teeth numbers 4 to 13 (maxillary right second premolar to maxillary left second premolar) sufficient to allow completion of the Study Dental Procedure. The maxillary teeth will be categorized in two subsets, anteriors (teeth numbers 6 to 11) and premolars (teeth numbers 4, 5, 12 and 13).

The intent is to treat 150 subjects at 3 study sites, 2:1 randomization within each study site, and an overall goal of 100 subjects treated with Kovacaine Mist and 50 treated with placebo. Recruitment will be from diverse dental patient populations with at least 25% of subjects over 50 years of age. Randomization will be within strata defined by age (≤50 and >50 years).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Need for an operative restorative dental procedure requiring local anesthesia for a single vital maxillary tooth (anterior or premolar tooth #4 to #13) with no evidence of pulpal pathology.
* Normal lip, nose, eyelid, and cheek sensation.
* Able to understand and sign the study informed consent document, communicate with the Investigators, and understand and comply with the requirements of the protocol.
* Patency of the naris ipsilateral to the tooth undergoing the Study Dental Procedure (the treatment tooth).
* Resting heart rate (HR) between 55 and 100 beats per minute (bpm), inclusive.
* Seated systolic blood pressure (SBP) between 95 and 150 mm Hg, inclusive, and seated diastolic blood pressure (DBP) between 60 and 100 mm Hg, inclusive.

Exclusion Criteria:

* Inadequately controlled hypertension (blood pressure greater than 150/100 mm Hg).
* Inadequately controlled active thyroid disease of any type.
* Frequent nose bleeds (≥ 5 per month).
* Having received dental care requiring a local anesthetic within the 24 hours preceding study entry.
* History of allergy to or intolerance of tetracaine, benzyl alcohol, other ester local anesthetics, or para-aminobenzoic acid (as found in PABA-containing sunscreen).
* History of allergy or hypersensitivity to articaine, oxymetazoline, epinephrine, or sulfite preservatives.
* Use of a monoamine oxidase inhibitor within the 3 weeks preceding study entry.
* Nursing, pregnant, suspected of being pregnant, or trying to become pregnant. (Females of child-bearing potential will be required to take a urine pregnancy test on the day of, but prior to, study drug administration to rule out pregnancy.)
* Having received any investigational drug and/or participation in any clinical trial within the 30 days prior to study participation.
* History of congenital or idiopathic methemoglobinemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Center for Dental Research Loma Linda University School, Loma Linda, California
  - University of Maryland, Baltimore, Baltimore, Maryland
  - University of Pennsylvania, School of Dental Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 3 sites in the U.S.
Groups:
- Kovacaine Mist: Tetracaine HCl 3% and Oxymetazoline HCl 0.05% - 2 sprays will be administered at the start of the procedure, if anesthesia is insufficient, a third spray will be administered.
  Tetracaine HCl 3% and Oxymetazoline HCl 0.05%
- Placebo: Placebo - 2 sprays will be administered at the start of the procedure, if anesthesia is insufficient, a third spray will be administered.
  Placebo
Period: Overall Study
Arm/Group | Kovacaine Mist | Placebo
Started | 100 | 50
Completed | 99 | 49
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovacaine Mist | Placebo | Total
Number analyzed (Participants) | 100 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (13.98) | 40.3 (15.23) | 41.2 (14.37)
Gender [Count of Participants; unit: Participants]
  Female | 57 | 25 | 82
  Male | 43 | 25 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 88 | 43 | 131
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 16 | 14 | 30
  Black or African American | 16 | 4 | 20
  White | 64 | 30 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 100 | 50 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic.
Description: If the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic and is considered a failure for this outcome.
Time Frame: at 15 minutes, +3 minute window
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 88 | 14

2. Secondary Outcome: Number of Participants Who Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic by Age Group (≤50 and >50 Years)
Description: If the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic and is considered a failure for this outcome. This outcome is broken down by age group, 1) less than 50 years of age and 2) 50 years of age and older.
Time Frame: at 15 minutes (+3 minute window) or 25 minutes (+3 minute window) if third intranasal spray is used
Population: Participants were only analyzed in their corresponding age group.
Measure: Number; unit: percentage of participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
percentage of participants
  less or = to 50: number analyzed (Participants) | 69 | 34
  less or = to 50 | 87 | 20.6
  greater than 50: number analyzed (Participants) | 31 | 16
  greater than 50 | 90.3 | 43.8

3. Secondary Outcome: Number of Participants With a Heart Rate Higher Than 125 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 0 | 0

4. Secondary Outcome: Number of Participants With a Heart Rate Lower Than 50 Bpm
Time Frame: at any time within 120 minutes following drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 4 | 1

5. Secondary Outcome: Number of Participants With an Increase From Baseline in Systolic Blood Pressure Greater Than or Equal to 25 mm Hg and/or to a Value Higher Than 160 mm Hg
Time Frame: at any time within 120 minutes following drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 5 | 2

6. Secondary Outcome: Number of Participants With a Decrease From Baseline in Systolic Blood Pressure Greater Than or Equal to 15 mm Hg and/or to a Value Lower Than 90 mm Hg
Time Frame: at any time within 120 minutes following study drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 1 | 1

7. Secondary Outcome: Number of Participants With an Increase From Baseline in Diastolic Blood Pressure Greater Than or Equal to 15 mm Hg and/or to a Value Higher Than 105 mm Hg
Time Frame: at any time within 120 minutes following study drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 1 | 1

8. Secondary Outcome: Number of Participants With a Decrease From Baseline in Diastolic Blood Pressure Greater Than or Equal to 10 mm Hg and/or to a Value Lower Than 50 mm Hg
Time Frame: at any time within 120 minutes following study drug administration
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
participants | 1 | 0

9. Secondary Outcome: Maximum Change From Baseline in Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
bpm | 5.3 (7.81) | 5.1 (9.02)

10. Secondary Outcome: Maximum Change From Baseline in Systolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
mmHg | 13.8 (10.18) | 9.2 (10.23)

11. Secondary Outcome: Maximum Change From Baseline in Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
mmHg | 11.1 (6.40) | 6.4 (6.53)

12. Secondary Outcome: The Profile Over Time of Heart Rate
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
beats per minute
  pre-study | 71.0 (10.37) | 73.6 (10.50)
  10 mins | 68.0 (10.66) | 72.6 (10.17)
  30 mins | 67.5 (10.86) | 66.3 (3.21)
  45 mins | 66.4 (10.52) | 70.9 (9.29)
  60 mins | 65.8 (10.26) | 69.2 (9.99)
  90 mins | 65.6 (10.27) | 67.7 (10.44)
  120 mins | 65.6 (9.65) | 68.9 (10.49)

13. Secondary Outcome: Alcohol Sniff Test
Description: The change from screening in the the distance from the nose (in centimeters) that a patient is able to detect the smell of alcohol on a cotton ball.
Time Frame: administered at approximately 24 hours after drug administration
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
cm | -0.8 (5.85) | 1.3 (6.17)

14. Secondary Outcome: The Profile Over Time of Systolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
mmHg
  pre-study | 123.1 (14.12) | 124.0 (13.70)
  10 mins | 128.6 (15.20) | 125.4 (16.02)
  30 mins | 117.3 (13.54) | 116.3 (10.26)
  45 mins | 125.0 (18.47) | 124.8 (18.27)
  60 mins | 127.1 (16.62) | 126.7 (18.79)
  90 mins | 128.8 (16.53) | 126.1 (15.89)
  120 mins | 129.5 (17.97) | 124.9 (15.54)

15. Secondary Outcome: The Profile Over Time of Diastolic Blood Pressure
Time Frame: from baseline to 120 minutes following drug administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 100 | 50
mmHg
  pre-study | 73.5 (9.37) | 74.7 (8.99)
  10 mins | 78.5 (10.64) | 75.2 (10.65)
  30 mins | 74.4 (9.13) | 67.0 (7.00)
  45 mins | 76.4 (10.50) | 74.7 (12.45)
  60 mins | 76.6 (10.71) | 76.7 (12.33)
  90 mins | 77.8 (10.53) | 75.4 (10.07)
  120 mins | 79.3 (10.75) | 75.4 (10.27)

16. Other Pre Specified Outcome: Number of Participants Who Received Three Sprays and Completed the Study Dental Procedure Without Need for Rescue by Injection of Local Anesthetic.
Description: A participant will receive two sprays and Study Dental Procedure will begin. If the participant does not have sufficient anesthesia a third sprays will be given. If after the third spray, the participant does not have sufficient anesthesia to complete the Study Dental Procedure, the participant is given a rescue injection of local anesthetic. This outcome analyzes just the participants who received the third spray and whether or not they completed the Study Dental Procedure without need for rescue by injection of local anesthesia.
Time Frame: at 25 minutes, +3 minute window
Population: This analysis is only of the participants who received 3 sprays. It does not include participants who only received 2 sprays.
Measure: Number; unit: participants
Arm/Group | Kovacaine Mist | Placebo
Number analyzed (Participants) | 27 | 33
participants | 16 | 0

ADVERSE EVENTS:
Time Frame: Approximately 24 hours following drug administration
Arm/Group | Kovacaine Mist | Placebo
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/50
Other Adverse Events (participants affected / at risk) | 83/100 | 15/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Kovacaine Mist (N=100) | Placebo (N=50)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 57 | 3 — (runny nose)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 27 | 3
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 24 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15 | 0 — (throat pain or discomfort)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 5 | 1 — (nasal stinging or burning sensation)
Dysgeusia (Nervous system disorders) | 7 | 1 — (abnormal taste sensation)
Headache (Nervous system disorders) | 9 | 1
Lacrimation Increased (Eye disorders) | 8 | 2 — (tearing or watery eyes)
Systolic BP Increased (Investigations) | 8 | 2
Diastolic BP Increased (Investigations) | 6 | 1
Intranasal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No